CLINICAL TRIAL: NCT05391945
Title: Effects of Thyroidectomy on Obstructive Sleep Apnea in Patients Suffering From Goiters
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: THYR_MB/AR/KP_2022
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Goiter
MeSH Terms: conditions — Goiter | interventions — Polysomnography; Respiratory Function Tests; Thyroid Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- goiter: Patients referred for partial/total thyroidectomy for goiter
  Interventions: Diagnostic Test: polysomnography

INTERVENTIONS:
Diagnostic Test: polysomnography — Patient will be assessed by home Polysomnography(PSG), one night, Pulmonary function tests, including respiratory muscle strength, and comprehensive biological assessment of thyroid function.
  Other Names: pulmonary function test; thyroid function tests

SUMMARY:
Literature regarding effects of goiter on the occurrence of obstructive sleep apnea (OSA) remains scarce. Reports have described cases of OSA in patients suffering from goiters, resolved after thyroidectomy.

It has been recently shown that goiters of a total volume exceeding 25 mL leads to >30% tracheal compression.

The aims of the present study is to assess 1) the prevalence of OSA in patients suffering from goiters and planned for thyroidectomy 2) the role of thyroidectomy in OSA resolution in patients suffering from pre-operative OSA 3) the identification of predictors for persisting OSA.

DETAILED DESCRIPTION:
Introduction

Literature regarding effects of goiter on the occurrence of obstructive sleep apnea (OSA) remains scarce. Reports have described cases of OSA in patients suffering from goiters, resolved after thyroidectomy.

It has been recently shown that goiters of a total volume exceeding 25 mL leads to >30% tracheal compression.

The aims of the present study is to assess 1) the prevalence of OSA in patients suffering from goiters and planned for partial/total thyroidectomy 2) the role of thyroidectomy in OSA resolution in patients suffering from pre-operative OSA 3) the identification of predictors for persisting OSA.

Methods

Design Prospective study Settings Tertiary referral center, university hospital Patients Patients referred for partial/total thyroidectomy for goiter Baseline assessment All patients planned for thyroidectomy will be prospectively included. Exclusion criteria will be: previous cervical surgery/radiotherapy, language barrier, chest disease known to narrow upper airways.

Patient will be assessed by home Polysomnography(PSG), one night, Pulmonary function tests, including respiratory muscle strength, and comprehensive biological assessment of thyroid function.

Follow up Three months after thyroidectomy, the same assessment will be repeated.

Statistical analysis

Statistical analysis will be performed to determine the percentage of patients suffering from OSA before surgery (apnea-hypopnea index (AHI) >5/hour of sleep on PSG). As the aim of the present study is to assess the role of thyroidectomy in OSA resolution, we will compare pre- and post-thyroidectomy PSG results in patients exhibiting AHI >5/hour of sleep (chi square test). OSA resolution will be defined as decrease in AHI > 50 % or reduction of AHI <5hour of sleep. As one of the secondary aim is the identification of predictors for persisting OSA, multivariate analysis will be performed to assess factors of persisting OSA, among age, neck circumference, body mass index, sex, pre/post menopausal status and pulmonary function tests parameters.

ELIGIBILITY:
Inclusion Criteria:

°patients planned for thyroidectomy for goiter

Exclusion Criteria:

* previous cervical surgery/radiotherapy
* language barrier
* chest disease known to narrow upper airways

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients planned for partial/total thyroidectomy for goiter
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
the prevalence of obstructive sleep apnea in patients suffering from goiters and planned for partial/total thyroidectomy | one month
  percentage

SECONDARY OUTCOMES:
OSA resolution after thyroidectomy in patients suffering from pre-operative OSA | three months after surgery
  percentage
body mass index is increased in patients with persisting OSA after surgery | three months after surgery
  weight and height will be combined to report BMI in kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No